CLINICAL TRIAL: NCT02375776
Title: Improving Outcomes in Cancer Patients on Oral Anti-Cancer Medications Using a Multi-modal mHealth Intervention
Brief Title: Improving Outcomes in Cancer Patients on Oral Anti-Cancer Medications Using a Multi-modal Mobile Health Intervention
Acronym: CORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McKesson Foundation (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-560.
Record Dates: First submitted 2014-12-24; First posted 2015-03-03 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Renal Cell Cancer; Prostate Cancer; Effects of Chemotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Download and use mobile health application - CORA- Device:smartphones for 12 weeks.
  Interventions: Other: CORA- Device:smartphones"
- Control (No Intervention): Usual Care - The control group will not use the study's mobile health application during the study.

INTERVENTIONS:
Other: CORA- Device:smartphones" — Participants will download and use Multi - modal mobile smartphone application (CORA -Device:smarthpones) designed for renal cell and prostate cancer patients taking anti-cancer medications
  Arms: Intervention

SUMMARY:
This study evaluates a smart phone based mobile application designed for patients with Renal Cell and Prostate Cancer taking oral anti-cancer medications. (OAMs) All participants will be patients at the Dana Farber Cancer Institute in Boston, Massachusetts. Half of the participants will use the mobile application for a 3 month period along with their usual care. Half of the participants will just receive usual care.

The investigators hope to show that cancer patients taking OAMs who use the mobile application will be better connected to their care team and will develop increased competency for self-care which will primarily increase medication adherence.

DETAILED DESCRIPTION:
The widespread and increasing use of oral anti-cancer medications (OAMs) has been ushered in by a rapidly increasing understanding of cancer pathophysiology. Furthermore, OAMs' popular ease of administration and potential cost savings has highlighted their central position in the healthcare system as a whole. Importantly, these facts have heightened appreciation of the unique challenges associated with OAMs use, especially in relation to prescribing, dispensing, reimbursement, education, adherence, and comprehensive quality and safety assurance. In this regard, the investigators goal is to improve medication adherence and clinical outcomes for cancer patients using OAMs through a mobile-enabled, multi-modal self-management and educational intervention .

The intervention seeks to enable patients' self-efficacy to adhere to their medications through directed education and coaching, anticipation of symptoms and associated adverse events, and closer monitoring with accurate assessment of self-reported outcomes. This innovative approach necessarily includes personalizing feedback and management based on patients' own treatment regimen, baseline knowledge and elucidated barriers to adherence, and holds great promise in improving overall adherence, safety, and clinical outcomes in these patients.

The investigators hypothesize that cancer patients on OAMs who use a mobile-based, multi-modal health self-management (M health) intervention designed for extensive patient education and symptom management will be better connected to their care team and will develop increased competency for self-care which will primarily increase medication adherence and improve secondary outcomes measured in this study compared to cancer patients on OAMs who do not use the mobile-based intervention.

ELIGIBILITY:
Inclusion Criteria:.

* Adult (≥18 years) patients being treated at the Dana Farber Cancer Institute for Renal Cell Cancer or Prostate Cancer commencing a new course cycle of OAMs. . - -Participants must be ambulatory and able to consent for self.
* Participants must have an Apple or Android smart phone and be willing to download the mobile application on their smartphones so they can utilize the intervention.
* Patients must be able to read/speak English.

Exclusion Criteria:

* Life expectancy less than 3 months as determined by the managing oncologist.
* Significant psychiatric co-morbidities and memory or cognitive impairments. A significant psychiatric condition includes any condition which creates major distress for a patient or which markedly impairs the patient's daily functioning. It includes, but not limited to, acute psychoses, major depressive disorder, dementia, etc
* Patients currently on similar interventional studies geared to improve medication adherence or in investigational drug trials in which adverse effects have not been fully elucidated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-03; Primary Completion 2018-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in Adherence to Oral Anti-Cancer Medications in patients with Renal Cell Cancer or Prostate Cancer on Oral Anti-Cancer Medications. | From randomization to end of study 12 weeks
  Medication adherence will be measured throughout the course of the study by the Medication Event Monitoring System. (Continuous data regarding medication adherence will be measured through this device and recorded in real time throughout the study - a period of 3 months.)

SECONDARY OUTCOMES:
Severity of symptoms in patients on Oral AntiCancer Medications. (OAMs) | From randomization to end of study 12 weeks
  Symptom severity will be measured using the MD Anderson Symptom Severity Inventory.
Hospital utilization in patients on OAMs. | From randomization to end of study 12 weeks
  Hospital utilization to include number of visits to Emergency Department visits, urgent clinic visits and in-patient admissions.
Quality of life metrics in patients on OAMs. | From randomization to end of study 12 weeks
  The Functional Assessment of Cancer Therapy-General (FACT-G) is an instrument used to measure health-related quality of life. been used extensively worldwide. The FACT-G has four subscales: Physical Well-Being (PWB), Social/Family Well-Being (SWB), Emotional Well-Being (EWB), and Functional Well-Being (FWB).
patient engagement with the mobile-based intervention in patients on OAMs. | From randomization to end of study 12 weeks
  Data will be collected for the 12 week duration of the study from the mobile application on participants' patterns of use of application. Additionally, Closeout Survey will asses user experience using the study mobile application and will collect user feedback.
Severity of anxiety in patients on OAMS. | From randomization to end of study 12 weeks
  The Generalized Anxiety Disorder 7 Item Scale GAD-7 will be used to screen for and assess severity of generalized anxiety disorder in patients using OAMS. The GAD-7 is a self-administered 7 question instrument. It is a valid and efficient tool to screen for and asses the severity of generalized anxiety disorder. It is used in both clinical practice and research.
Severity of fatigue in patients on OAMs. | From randomization to end of study 12 weeks
  The Functional Assessment of Chronic Illness Therapy - Fatigue Version (FACIT-F) will be used to assess patient fatigue. It is a self administered 13 question instrument validated for use in chronic illness and frequently used with cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Jethwani, MD, MPH, Principal Investigator — Center for Connected Health, Partners HealthCare
Locations (1):
- Partners HealthCare Connected Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided